CLINICAL TRIAL: NCT02411877
Title: REperfusion With Cooling in CerebraL Acute IscheMia II
Acronym: RECCLAIM-II
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: It was decided that it was not feasible to continue this study.
Sponsor: WellStar Health System (Other)
Collaborators: Zoll Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RECCLAIM II-S
Record Dates: First submitted 2015-03-25; First posted 2015-04-08 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Ischemic Stroke; Hypothermia
Keywords: Acute ischemic stroke; Mild hypothermia; Stroke; Hypothermia; Cerebral infarction; Ischemia; Cerebrovascular disorder; Brain disease; Central nervous system disease; Nervous system disease; Vascular disease; Cardiovascular disease; Brain infarction; Brain ischemia; Pathologic process; Body temperature change; Signs and symptoms
MeSH Terms: conditions — Ischemic Stroke; Hypothermia; Stroke; Cerebral Infarction; Ischemia; Cerebrovascular Disorders; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Vascular Diseases; Cardiovascular Diseases; Brain Infarction; Brain Ischemia; Pathologic Processes; Body Temperature Changes; Signs and Symptoms | interventions — Reperfusion; Hypothermia, Induced

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normothermia (Active Comparator): As part of standard of care, an interventional reperfusion procedure will be performed on all subjects using the Trevo Pro Retriever (Stryker), after which normothermia will attempt to keep core body temp between 38 and 36.5 degrees centigrade.
  Interventions: Procedure: Normothermia; Device: Trevo Pro Retriever (Stryker Corp.)
- Mild hypothermia (Experimental): As part of standard of care, an interventional reperfusion procedure will be performed on all subjects using the Trevo Pro Retriever (Stryker). Subjects will also have a catheter placed in the femoral vein (Zoll Thermogard XP technology with the Quattro catheter) and temperature brought to 33 degrees centigrade as quickly as possible. They will stay in mild hypothermia for 12 hours, and then be rewarmed very slowly.
  Interventions: Procedure: Mild hypothermia; Device: Trevo Pro Retriever (Stryker Corp.); Device: Zoll Thermogard XP technology with the Quattro catheter

INTERVENTIONS:
Procedure: Normothermia — Device: Trevo Pro Retriever (Stryker Corp.)
  Other Names: Clot retrieval, reperfusion
  Arms: Normothermia
Procedure: Mild hypothermia — Device: Zoll Thermogard XP technology with the Quattro catheter Device: Trevo Pro Retriever (Stryker Corp.)
  Other Names: Therapeutic hypothermia, clot retrieval, reperfusion
  Arms: Mild hypothermia
Device: Trevo Pro Retriever (Stryker Corp.) — Device: Trevo Pro Retriever (Stryker Corp.)
Device: Zoll Thermogard XP technology with the Quattro catheter — Device: Zoll Thermogard XP technology with the Quattro catheter
  Arms: Mild hypothermia

SUMMARY:
The purpose of this study is to determine whether reducing a patient's body temperature (mild hypothermia of 33 degrees Centigrade) will significantly reduce the risk of brain injury (notably reperfusion injury and hemorrhagic conversion) in patients who have suffered a significant interruption of blood flow to an area of brain (occlusion of large proximal cerebral artery) and have undergone successful removal of that interruption (revascularization).This will be achieved by comparing patients who have undergone hypothermia to those who have not.

DETAILED DESCRIPTION:
This study is designed to examine the safety and proof of concept of therapeutic hypothermia prior to conventional revascularization in subjects experiencing acute ischemic stroke by comparing the results to subjects who remain at normal body temperature (normothermic) and proceed directly to reperfusion via conventional reperfusion intervention.

The investigational plan also examines the following outcomes in 85 subjects randomized to either hypothermia or normothermia:

* Regulation of biomarkers indicative of ischemia-reperfusion injury
* Changes in blood brain injury using the Hyperintense Acute Reperfusion Marker (HARM) protocol MRI as a surrogate imaging biomarker
* Incidence of hemorrhagic conversion post reperfusion
* Neurologic function at 90 days post acute ischemic stroke.

The results of this study will be used to power a definitive phase III clinical trial evaluating the combination of hypothermia and revascularization versus reperfusion alone.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects of any ethnicity and age >/=18 but </= 79 years;
* Symptom onset </=8 hours;
* Symptoms consistent with an ischemic stroke with a large vessel occlusion (Middle Cerebral Artery (MCA), Internal Carotid Artery (ICA) terminus) as determined by CT imaging of the brain;
* Alberta Stroke Program Early CT Score (ASPECTS) of 5-10 on non-contrast CT of the brain;
* Ability to undergo endovascular reperfusion therapy;
* No contraindications to general anesthesia, conscious sedation, or allergies to any components associated with the anticipated diagnostic or treatment procedures that cannot be treated;
* A pre-treatment modified Rankin Scale (mRS) of 0 or 1;
* Baseline CT scan shows no hemorrhage;
* National Institutes of Health Stroke Scale (NIHSS) 14-29;
* Subject has either 1) failed iv tissue plasminogen activator (tPA) therapy or 2) contradicted for iv tPA therapy;
* Subject is capable of complying with study procedures and agrees to complete all required study procedures, study visits and associated activities.
* Subject or legally authorized representative must be able to understand and give written informed consent.

Exclusion Criteria:

* Females of childbearing potential who are pregnant or not using adequate contraception;
* Bleeding diathesis with a platelet count < 50,000 or International Normalized Ratio (INR) >1.7 or any active or recent (within 10 to 30 days) hemorrhage;
* History of genetically confirmed hypercoagulable syndrome;
* Any condition that excludes MRI imaging;
* History of dementia, currently on Aricept or Namenda, or other Alzheimer's-like symptoms;
* End stage renal disease on hemodialysis;
* History of cardiac arrest;
* Presence of an inferior vena cava (IVC) filter;
* Contrast dye allergy with history of anaphylaxis, known serious sensitivity to contrast agents or any condition in which angiography is contraindicated;
* Known allergy to meperidine or buspar;
* Prior neurologic event that would obscure interpretation of the signal and current presenting neurologic deficits;
* Sustained hypertension (systolic blood pressure (SBP) > 185 or diastolic blood pressure (DBP) > 110 refractory to treatment);
* Baseline CT/MRI of head showing evidence of mass effect with mid-line shift, hemorrhage, intracranial tumor, arterial vasculitis or dissection, or bilateral stroke;
* Presence of any other serious comorbidity that would be likely to impact life expectancy to less than 6 months or limit subject cooperation or study compliance;
* Concurrent participation in an investigational clinical study that has not completed the follow-up period or planned participation in another study within the next 3 months;
* Any other condition or personal circumstance that, in the judgment of the investigator, might interfere with the collection of complete, good quality data or the completion of the research study.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-02; Primary Completion 2017-11 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
Hemorrhagic Conversion | 48 hours
  Acute bleeding into the area of the original stroke based on CT or MRI of the head.

SECONDARY OUTCOMES:
Hyperintense Acute Reperfusion Marker (HARM) | 48 +/- 24 hours
  HARM is a MRI sequence looking at gadolinium enhancement on FLAIR MRI imaging.
National Institutes of Health Stroke Scale (NIHSS) | Baseline, 24 +/- 6 hours, 48 +/- 24 hours, 8 +/- 2 days, 90 +/- 15 days
  NIHSS is a scale from 1-42 to evaluate stroke severity
Modified Rankin Scale (mRS) | Basline, 48 +/- 24 hours, 90 +/- 15 days
  mRS is a straightforward evaluation of the functional limitations from stroke
Number of participants with adverse events | 90 days
  Evaluation and determination of the following complications pneumonias, central line infections, intra-cerebral hemorrhages, systemic hemorrhages, transient cerebral ischemia, and new strokes.

CONTACTS AND LOCATIONS:
Overall Officials: Rishi Gupta, MD, Study Director — WellStar Health System
Locations (1):
- WellStar Kennestone Regional Medical Center, Marietta, Georgia, United States